CLINICAL TRIAL: NCT03921489
Title: Subchondroplasty for Treatment of Bone Marrow Edema in the Foot and Ankle
Status: Completed | Type: Observational
Sponsor: Ellianne M. Nasser (Other)
Responsible Party: Sponsor-Investigator, Ellianne M. Nasser, Staff Physician, Geisinger Clinic
Organization: Geisinger Clinic (Other)
Other Study IDs: 2019-0221
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-09

CONDITIONS: Bone Marrow Edema
Keywords: bone marrow edema; subchondroplasty; foot and ankle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subchondroplasty in treating bone marrow edema: These patients will have calcium phosphate mineral compound injected into the bone marrow lesions.
  Interventions: Procedure: Subchondroplasty

INTERVENTIONS:
Procedure: Subchondroplasty — Calcium phosphate mineral compound injected into the bone marrow lesions

SUMMARY:
The subchondroplasty procedure has been used to treat bone marrow edema mostly located in the periarticular region of the knee. In the past few years, it has expanded its use in the foot and ankle. There has, however, been very minimal research documented on its utilization in that area. This study aims to prospectively evaluate the course of treatment and outcomes of painful bone marrow lesions in these associated podiatric circumstances using subchondroplasty. It is hypothesized that use of calcium phosphate bone substitute in the foot and ankle to treat bone marrow edema will have more favorable short and long-term outcomes than joint destructive and joint sparing procedures more commonly performed for treatment in the past.

DETAILED DESCRIPTION:
The subchondroplasty procedure has been used to treat bone marrow edema mostly located in the periarticular region of the knee. In the past few years, it has expanded its use in the foot and ankle. There has, however, been very minimal research documented on its utilization in that area. Bone marrow edema arises from altered stresses on bones due to osteoarthritis, biomechanical abnormalities, coalitions, infection, and trauma. This study aims to prospectively evaluate the course of treatment and outcomes of painful bone marrow lesions in these associated podiatric circumstances using subchondroplasty. This should, therefore, expose this modality as a viable treatment option for bone marrow edema.

Patients will be evaluated in the office/clinic setting with a positive diagnosis of bone marrow edema confirmed via MRI. They must have failed 3 months of conservative treatment measures including, but not limited to, orthotic modifications, taping, immobilization or offloading, and anti-inflammatories. The study population includes individuals over the age of 18 with no significant comorbidities or previous foot and ankle surgical interventions. These patients will go on to have calcium phosphate mineral compound injected into the bone marrow lesions. We will track the progression of their symptoms and evaluate via Visual Analog Scale (VAS) pain score and the American Orthopedic Foot and Ankle Score (AOFAS) at 3-month, 6-month, and 1-year follow-ups.

The subchondroplasty procedure is a viable treatment option for bone marrow edema in the setting of altered pedal biomechanics, gait abnormalities, osteoarthritis, and trauma. It is a minimally invasive procedure that maximizes positive outcomes, allows the patient to be immediately weight bearing following surgery, and has short operating room times. This surgical procedure is a new and innovative technique introduced to the podiatric field that will allow the surgeon to intervene at an earlier stage in efforts to alleviate symptoms. It is hypothesized that use of calcium phosphate bone substitute in the foot and ankle to treat bone marrow edema will have more favorable short and long-term outcomes than joint destructive and joint sparing procedures more commonly performed for treatment in the past.

ELIGIBILITY:
Inclusion Criteria:

* Bone marrow edema diagnosed on MRI
* Pain in the foot and ankle due to the presence of bone marrow edema
* Failed 3 months of conservative treatment

Exclusion Criteria:

* Patient <18 years of age
* Presence of osteomyelitis of poor surgical candidates due to comorbidities such as diabetics with an HbA1c of >8%
* Patient with previous foot and ankle surgeries that may interfere with future outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bone marrow edema diagnosed on MRI who elect to receive subchondroplasty procedure
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for pain | 0-12 months
  Best 0-10 worst - Continuous scale to measure current pain level
Subchondroplasty Patient Satisfaction Survey | 0-12 months
  Worst 0-5 best. 5-item scale to measure patient satisfaction after subchondroplasty procedure
The American Orthopedic Foot and Ankle Score (AOFAS) | 0-12 months
  Worst 0-100 best

CONTACTS AND LOCATIONS:
Overall Officials: Ellianne Nasser, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Community Medical Center, Scranton, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No